CLINICAL TRIAL: NCT00924170
Title: Phase II Trial of LMB-2, Fludarabine and Cyclophosphamide for Adult T-Cell Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Kreitman, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090025; 09-C-0025; NCT00794833 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Adult T-Cell Leukemia (ATL)
Keywords: Immunotoxin; CD25; Immunogenicity; Neutralization; Neutralizing Antibodies; Adult T-Cell Leukemia; Leukemia; ATL
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell; Leukemia | interventions — B3(Fv)-PE38KDEL recombinant immunotoxin; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine and Cyclophosphamide/LMB-2 (Experimental): Administer cycle 1 with Fludarabine and Cyclophosphamide (FC) alone. Two weeks after starting cycle 1, begin up to 6 cycles of FC plus LMB-2 at minimum 20-day intervals.
  Interventions: Drug: LMB-2; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: LMB-2 — Begin with 30 mcg/Kg intravenous (IV) on days 3, 5 and 7. Escalate to 40 mcg/Kg if dose limiting toxicity (DLT) in 0/3 or 1/6 at 30 mcg/Kg. Continue at 40 mcg/Kg if 0-1 of 6 have DLT at 40 mcg/Kg.
Drug: Fludarabine — Days 1-3:
  Patients 1-7, 10-14, and >18:25mg/m^2/day Patients 8 - 9:30 mg/m^2/day Patients 15- 17:20 mg/m^2/day
  Other Names: Fludara
Drug: Cyclophosphamide — Days 1-3:
  Patients 1-7, 10 -14, and >18:250 mg/m^2/day Patients 8 - 9:300 mg/m^2/day Patients 15-17:200 mg/m^2/day
  Other Names: Cytoxan

SUMMARY:
BACKGROUND:

* Cluster of differentiation 25 (CD25) (p55, Tac or interleukin 2 receptor (IL2R) alpha) is strongly expressed in virtually 100% of patients with adult T-cell leukemia/lymphoma (ATL), a highly aggressive human T-lymphotropic virus type 1 (HTLV-1) related malignancy responding poorly to chemotherapy.
* In ATL, the humanized anti-CD25 monoclonal antibody (Mab) daclizumab produced 13-14% responses, and the anti-CD52 Mab Alemtuzumab (Campath-1H) produced response lasting greater than 2 months in 30% of 23 patients.
* LMB-2 is an anti-CD25 recombinant immunotoxin containing variable domains of murine MAb anti-Tac and truncated Pseudomonas exotoxin.
* In a phase I trial at National Cancer Institute (NCI), the maximum tolerated dose (MTD) of LMB-2 was 40 microg/Kg intravenous (IV) given every other day for 3 doses (every other day (QOD) times 3). LMB-2 induced greater than 90% tumor reduction rapidly in all 3 ATL patients on protocol, but achieved only 1 partial response due to rapid tumor progression and/or immunogenicity.
* In preclinical models, response from recombinant immunotoxins is limited by high concentrations of soluble receptor in the blood and especially in the interstitial space of the tumor. Synergism was observed with chemotherapy and immunotoxins, possibly due to reduction of soluble receptor in tumor interstitium.

OBJECTIVES:

-To determine, in nonrandomized fashion, if after verifying its safety, fludarabine and cyclophosphamide (FC) prior to LMB2 for ATL can result in low immunogenicity and a rate of major response lasting greater than 2 months, which may be an improvement over that demonstrated previously from Alemtuzumab (CAMPATH).

Secondary objectives:

* To determine the effect of 1 cycle of FC alone in ATL.
* To examine progression-free and overall survival in ATL after FC/LMB-2.
* Evaluate pharmacokinetics, toxicity, and monitor soluble CD25 and other tumor marker levels in the serum.
* To study the effects of LMB-2 plus FC on normal B- and T-cell subsets by fluorescence-activated cell sorting (FACS).

ELIGIBILITY:

* CD25 plus ATL, untreated or with prior therapy
* Eastern Cooperative Oncology Group (ECOG) 0-2, absolute neutrophil count (ANC), platelets and albumin at least 1000, 75,000, and 3.0.

DESIGN:

* Fludarabine 25 mg/m(2) IV days 1-3
* Cyclophosphamide 250 mg/m(2) IV days 1-3
* LMB-2 30-40 micro g/Kg IV days 3, 5 and 7.
* LMB-2 dose: Begin with 30 microg/Kg times 3. Escalate to 40 microg/Kg if dose limiting toxicity (DLT) in 0/3 or 1/6 at 30 microg/Kg. Continue at 40 microg/Kg if 0-1 of 6 have DLT at 40 microg/Kg.
* Administer cycle 1 with FC alone. Two weeks after starting cycle 1, begin up to 6 cycles of FC plus LMB-2 at minimum 20-day intervals.
* Accrual goals: 29-37 patients, which includes 4 replacements....

DETAILED DESCRIPTION:
BACKGROUND:

* Cluster of differentiation 25 (CD25) (p55, Tac or interleukin receptor 2 (IL2Ra) is strongly expressed in virtually 100 % of patients with adult T-cell leukemia/lymphoma (ATL), a highly aggressive human T-lymphotropic virus type 1 (HTLV-1) related malignancy responding poorly to chemotherapy.
* In adult T-cell leukemia (ATL), the humanized anti-CD25 monoclonal antibody (Mab) daclizumab produced 13-14 % responses, and the anti-CD52 Mab Alemtuzumab (Campath- 1H) produced response lasting > 8 weeks in of 30 % of 23 patients.
* LMB-2 is an anti-CD25 recombinant immunotoxin containing variable domains of murine MAb anti-Tac and truncated Pseudomonas exotoxin.
* In a phase I trial at National Cancer Institute (NCI), the maximum tolerated dose (MTD) of LMB-2 was 40 mcg/Kg dose intravenous (IV) given every other day for 3 doses (every other day (QOD) x3). LMB-2 induced > 90 % tumor reduction rapidly in all 3 ATL patients on protocol, but achieved only 1 partial response due to rapid tumor progression and/or immunogenicity.
* In preclinical models, response from recombinant immunotoxins is limited by high concentrations of soluble receptor in the blood and especially in the interstitial space of the tumor. Synergism was observed with chemotherapy and immunotoxins, possibly due reduction of soluble receptor in tumor interstitium.

OBJECTIVES:

* To determine, in nonrandomized fashion, if after verifying its safety, fludarabine and cyclophosphamide (FC) prior to LMB2 for ATL can result in low immunogenicity and a rate of major response lasting > 8 weeks which may be an improvement over that demonstrated previously from Alemtuzumab (CAMPATH).
* Secondary objectives

  * To determine the effect of 1 cycle of FC alone in ATL.
  * To examine progression-free and overall survival in ATL after FC/LMB-2.
  * Evaluate pharmacokinetics, toxicity, and monitor soluble CD25 and other tumor marker levels in the serum.
  * To study the effects of LMB-2 +FC on normal B- and T-cell subsets by FACS.

ELIGIBILITY:

* CD25+ ATL, untreated or with prior therapy, leukemic type without malignant masses > 4 cm.
* Eastern Cooperative Oncology Group (ECOG) 0-2, absolute neutrophil count (ANC), platelets and albumin at least 1000, 75,000, and 3.0 respectively.

DESIGN:

* IV fludarabine and cyclophosphamide (FC) days 1-3 (doses listed respectively)
* Patients 1-7 and 10-14, and >18: 25 and 250 mg/m^2/day
* Patients 8-9: 30 and 300 mg/m^2/day
* Patients 15-17: 20 and 200 mg/m^2/day
* LMB-2 dose: Begin with 30 mcg/Kg IV on days 3,5 and 7. Escalate to 40 mcg/Kg if dose limiting toxicity (DLT) in 0/3 or 1/6 at 30 mcg/Kg. Continue at 40 mcg/Kg if 0-1 of 6 have DLT at 40 mcg/Kg.
* Administer cycle 1 with FC alone. Two weeks after starting cycle 1, begin up to 6 cycles of FC plus LMB-2 at minimum 20 day intervals.
* Accrual goals: 29-37 patients, which includes 4 replacements.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis of acute or lymphomatous adult T-cell leukemia (ATL) by flow cytometry of blood or immunohistochemistry of biopsy tissue, confirmed by National Cancer Institute (NCI) Laboratory of Pathology, and previously treated unless the patient is ineligible for or refuses other protocols or treatments for ATL.
  2. Neutralizing antibodies less than or equal to 75% neutralization of 200 ng/ml of LMB-2.
  3. At least 18 years old.
  4. Eastern Cooperative Oncology Group (ECOG) 0-2.
  5. Able to understand and give informed consent.
  6. Negative pregnancy test for females of childbearing potential.
  7. The transaminases alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must each be less than or equal to 3-times the upper limits of normal (UNL) or less than or equal to 10-times normal if due to ATL. Albumin must be greater than or equal to 3.0 gm/dL. Total bilirubin must be less than or equal to 1.5 mg/dL except in patients with Gilberts syndrome (as defined by greater than 80 percent unconjugated bilirubin) it must be less than 5mg/dl.
  8. Creatinine less than 2.0 mg/dL.
  9. Absolute neutrophil count (ANC) greater than or equal to 1000/uL and platelets greater than or equal to 50,000/uL.
  10. Current or prior features of acute ( corrected calcium (Ca)++ > 2.73 or lactate dehydrogenase (LDH) 2- fold above ULN) or chronic (LDH 1.5-2-fold above ULN or absolute lymphocyte count >4 x10^9/L with T-cells >3.5 x10^9/L) ATL. Patients with smoldering ATL (no acute or chronic features) and symptomatic ATL skin lesions are also eligible.

EXCLUSION CRITERIA:

1. Prior therapy with LMB-2.
2. Central nervous system disease as evidenced by clinical symptomatology.
3. Cytotoxic chemotherapy, steroids or monoclonal antibody (Mab) within 3 weeks of enrollment, except anti Tac Mab (i.e. daclizumab), which cannot be used within 12 weeks of enrollment. Hydroxyurea is considered different from cytotoxic chemotherapy and may be used up to the day before enrollment providing it is not increased during the week prior to enrollment and that patients disease burden is not decreasing during that time.
4. Uncontrolled infection.
5. Untreated or uncontrolled 2nd malignancy.
6. Patients who are pregnant or breast-feeding.
7. Patients who have human immunodeficiency virus (HIV) or hepatitis C, since in these patients reductions in normal T- or B-cells would increase the risk of exacerbation of their underlying disease. Patients would not be excluded for hepatitis B surface antigen positivity if on Lamivudine or Entecavir.
8. Patients receiving warfarin (Coumadin [R])
9. Patients with a left ventricular ejection fraction of less than 45%.
10. Patients with a diffusing capacity of the lungs for carbon monoxide (DLCO) less than 50% of normal or an forced expiratory volume 1 (FEV1) less than 50% of normal.
11. No concomitant use of alternative complimentary therapies or over the counter (OTC) agents allowed without prior approval of the principal investigator (PI).
12. Tumor or lymph node masses > 4 cm.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10-31 (Actual); Primary Completion 2016-01-02 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Waldmann TA, Greene WC, Sarin PS, Saxinger C, Blayney DW, Blattner WA, Goldman CK, Bongiovanni K, Sharrow S, Depper JM, et al. Functional and phenotypic comparison of human T cell leukemia/lymphoma virus positive adult T cell leukemia with human T cell leukemia/lymphoma virus negative Sezary leukemia, and their distinction using anti-Tac. Monoclonal antibody identifying the human receptor for T cell growth factor. J Clin Invest. 1984 Jun;73(6):1711-8. doi: 10.1172/JCI111379. PMID 6327770
- [Background] Leonard WJ, Depper JM, Uchiyama T, Smith KA, Waldmann TA, Greene WC. A monoclonal antibody that appears to recognize the receptor for human T-cell growth factor; partial characterization of the receptor. Nature. 1982 Nov 18;300(5889):267-9. doi: 10.1038/300267a0. No abstract available. PMID 6815536
- [Background] Proietti FA, Carneiro-Proietti AB, Catalan-Soares BC, Murphy EL. Global epidemiology of HTLV-I infection and associated diseases. Oncogene. 2005 Sep 5;24(39):6058-68. doi: 10.1038/sj.onc.1208968. PMID 16155612
- [Background] Kreitman RJ, Stetler-Stevenson M, Jaffe ES, Conlon KC, Steinberg SM, Wilson W, Waldmann TA, Pastan I. Complete Remissions of Adult T-cell Leukemia with Anti-CD25 Recombinant Immunotoxin LMB-2 and Chemotherapy to Block Immunogenicity. Clin Cancer Res. 2016 Jan 15;22(2):310-8. doi: 10.1158/1078-0432.CCR-15-1412. Epub 2015 Sep 8. PMID 26350263
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0025.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC: Leukemic patients receiving LMB-2 and at least 25+250 mg/m^2 fludarabine and cyclophosphamide; CF03-CF05, CF07-CF10, and CF12-CF14.
- All Other Patients: Patients CF01-CF02, CF06, CF11, and CF15-CF18. This is a mixture of patients who did not receive LMB-2, who had lymphoma-type adult T-cell leukemia, and who received 20+250 mg/m^2 of fludarabine cyclophosphamide (FC).
Period: Overall Study
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Started | 10 | 8
Completed | 3 | 0
Not Completed | 7 | 8
Not completed — Refused further treatment | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Progressive disease | 3 | 6
Not completed — Stopped due to neutralizing antibodies | 3 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14.25) | 39.8 (10.77) | 40.9 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 2 | 2 | 4
  Tabago, Black | 1 | 0 | 1
  Peruvian, Hispanic | 1 | 0 | 1
  American from Jamaica, Black | 1 | 0 | 1
  Jamaican, Black | 5 | 2 | 7
  Ethiopian, Black | 0 | 1 | 1
  Jamaican | 0 | 0 | 0
  Barbados, Black | 0 | 2 | 2
  American, from Ghana, Black | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 18
Prior Treatment [Count of Participants; unit: Participants] — Prior treatments included cyclophosphamide, adriamycin, vincristine, and prednisone (CHOP), these 4 agents with etoposide (EPOCH) and campath (C or alemtuzumab, together EPOCH-C), etoposide, methylprednisolone, cytarabine, and cisplatin (ESHAP), pralatrexate (PTX), gemcitabine (Gem), siplizumab (Medi507), denileukin diftitox (Ontak), daclizumab or humanized anti-Tac (HAT) and EPOCH with rituximab and siplizumab (EPOCH-RS). The LSG-15 regimen includes prednisone, adriamycin, carmustine, etoposide, carboplatin, and vinorelbine. Population: One participant was not evaluable. Participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2.
  Participants
    CHOP: number analyzed (Participants) | 10 | 7 | 17
    CHOP | 2 | 3 | 5
    EPOCH-C: number analyzed (Participants) | 10 | 7 | 17
    EPOCH-C | 0 | 1 | 1
    C, ESHAP, PTX, Gem: number analyzed (Participants) | 10 | 7 | 17
    C, ESHAP, PTX, Gem | 1 | 0 | 1
    Medi507, Ontak, HAT: number analyzed (Participants) | 10 | 7 | 17
    Medi507, Ontak, HAT | 1 | 0 | 1
    CHOP, C: number analyzed (Participants) | 10 | 7 | 17
    CHOP, C | 2 | 0 | 2
    EPOCH-RS: number analyzed (Participants) | 10 | 7 | 17
    EPOCH-RS | 1 | 1 | 2
    None: number analyzed (Participants) | 10 | 7 | 17
    None | 1 | 0 | 1
    Hydroxyurea: number analyzed (Participants) | 10 | 7 | 17
    Hydroxyurea | 1 | 1 | 2
    CHOP, Hydroxyurea: number analyzed (Participants) | 10 | 7 | 17
    CHOP, Hydroxyurea | 1 | 0 | 1
    LSG-15, radiation: number analyzed (Participants) | 10 | 7 | 17
    LSG-15, radiation | 0 | 1 | 1
Type of Leukemia [Count of Participants; unit: Participants] — Population: One participant was not evaluable. Participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2.
  Participants
    Acute: number analyzed (Participants) | 10 | 7 | 17
    Acute | 10 | 3 | 13
    Lymphoma: number analyzed (Participants) | 10 | 7 | 17
    Lymphoma | 0 | 4 | 4
Extravascular sites [Count of Participants; unit: Participants] — Population: One participant was not evaluable. Participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2.
  Participants
    Bone, lung, skin: number analyzed (Participants) | 10 | 7 | 17
    Bone, lung, skin | 0 | 1 | 1
    Thigh (skin): number analyzed (Participants) | 10 | 7 | 17
    Thigh (skin) | 0 | 1 | 1
    Pelvis: number analyzed (Participants) | 10 | 7 | 17
    Pelvis | 1 | 0 | 1
    Muscle: number analyzed (Participants) | 10 | 7 | 17
    Muscle | 1 | 0 | 1
    Skin: number analyzed (Participants) | 10 | 7 | 17
    Skin | 1 | 0 | 1
    Lymph node (LN): number analyzed (Participants) | 10 | 7 | 17
    Lymph node (LN) | 1 | 2 | 3
    Spleen, LN: number analyzed (Participants) | 10 | 7 | 17
    Spleen, LN | 2 | 1 | 3
    Subcutaneous: number analyzed (Participants) | 10 | 7 | 17
    Subcutaneous | 1 | 1 | 2
    None: number analyzed (Participants) | 10 | 7 | 17
    None | 1 | 0 | 1
    Bone, subcutaneous: number analyzed (Participants) | 10 | 7 | 17
    Bone, subcutaneous | 0 | 1 | 1
    Spleen: number analyzed (Participants) | 10 | 7 | 17
    Spleen | 2 | 0 | 2
Participants with High Lactate Hydrogenase (LDH) [Count of Participants; unit: Participants] — High LDH is > 400 u/L. Population: One participant was not evaluable. Participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2.
  Participants
    Yes: number analyzed (Participants) | 10 | 7 | 17
    Yes | 10 | 7 | 17
    No: number analyzed (Participants) | 10 | 7 | 17
    No | 0 | 0 | 0
Participants with High Calcium++ [Count of Participants; unit: Participants] — High Calcium++ is a corrected calcium > 2.74 Population: One participant was not evaluable. Participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2.
  Participants
    Yes: number analyzed (Participants) | 10 | 7 | 17
    Yes | 5 | 2 | 7
    No: number analyzed (Participants) | 10 | 7 | 17
    No | 5 | 5 | 10
Adult T-cell Leukemia (ATL) cells/mm^3 in the Peripheral Blood [Count of Participants; unit: Participants] — Population: One participant was not evaluable. Participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2.
  Participants
    0 cells: number analyzed (Participants) | 10 | 7 | 17
    0 cells | 0 | 3 | 3
    1 cell: number analyzed (Participants) | 10 | 7 | 17
    1 cell | 0 | 1 | 1
    80 cells: number analyzed (Participants) | 10 | 7 | 17
    80 cells | 1 | 0 | 1
    206 cells: number analyzed (Participants) | 10 | 7 | 17
    206 cells | 1 | 0 | 1
    246 cells: number analyzed (Participants) | 10 | 7 | 17
    246 cells | 1 | 0 | 1
    408 cells: number analyzed (Participants) | 10 | 7 | 17
    408 cells | 1 | 0 | 1
    450 cells: number analyzed (Participants) | 10 | 7 | 17
    450 cells | 0 | 1 | 1
    687 cells: number analyzed (Participants) | 10 | 7 | 17
    687 cells | 1 | 0 | 1
    5,604 cells: number analyzed (Participants) | 10 | 7 | 17
    5,604 cells | 1 | 0 | 1
    7,737 cells | 0 | 1 | 1
    8,216 cells: number analyzed (Participants) | 10 | 7 | 17
    8,216 cells | 1 | 0 | 1
    13,153 cells: number analyzed (Participants) | 10 | 7 | 17
    13,153 cells | 1 | 0 | 1
    24,112 cells: number analyzed (Participants) | 10 | 7 | 17
    24,112 cells | 1 | 0 | 1
    210,000 cells: number analyzed (Participants) | 10 | 7 | 17
    210,000 cells | 1 | 0 | 1
    213,000 cells: number analyzed (Participants) | 10 | 7 | 17
    213,000 cells | 0 | 1 | 1
Maximum tumor size [Count of Participants; unit: Participants] — Maximum tumor size is listed, respectively, with the maximum spleen diameter. Population: One participant was not evaluable. Participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2.
  Participants
    <1 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    <1 cm tumor | 4 | 1 | 5
    1.9 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    1.9 cm tumor | 0 | 1 | 1
    2 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    2 cm tumor | 1 | 0 | 1
    2.2 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    2.2 cm tumor | 0 | 1 | 1
    5.6 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    5.6 cm tumor | 1 | 0 | 1
    5.8 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    5.8 cm tumor | 0 | 1 | 1
    6 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    6 cm tumor | 0 | 1 | 1
    9 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    9 cm tumor | 0 | 1 | 1
    15, 2.5 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    15, 2.5 cm tumor | 0 | 1 | 1
    17 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    17 cm tumor | 1 | 0 | 1
    17.5 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    17.5 cm tumor | 1 | 0 | 1
    18.5, 1.7 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    18.5, 1.7 cm tumor | 1 | 0 | 1
    20, 1.8 cm tumor: number analyzed (Participants) | 10 | 7 | 17
    20, 1.8 cm tumor | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Minimally Durable Clinical Response Rate
Description: Response is based on the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma and must last >8 weeks to meet the primary endpoint of the study. Complete remission (CR) is complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related symptoms if present before therapy and normalization of those biochemical abnormalities definitely assignable to the lymphoma. Partial response is reduction by ≥50% of leukemia cell count or ≥50% reduction in the size of all measurable lesions, and no increase in size of any measurable or evaluable lesion or appearance of new lesion. Stable disease is neither a response nor progressive disease. Progressive disease is appearance of new lesions, or an increase of 50% or greater in the sum of the product of the perpendicular diameters of the measurable lesions or persistent (at least two determinations) doubling of the peripheral blood leukemic cell count.
Time Frame: 8 weeks
Population: All 10 patients receiving LMB-2 and at least 25+250 mg/m^2 Fludarabine/Cyclophosphamide (FC) were evaluable for response.
  Of the 8 other patients, only 5 received LMB-2 and were therefore evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 8
percentage of participants
  Overall Response: number analyzed (Participants) | 10 | 5
  Overall Response | 80 [44.4 to 97.5] | 0 [0 to 0]
  Complete Response: number analyzed (Participants) | 10 | 5
  Complete Response | 60 [26 to 88] | 0 [0 to 0]
  Partial Response: number analyzed (Participants) | 10 | 5
  Partial Response | 20 [2.5 to 55.6] | 0 [0 to 0]
  Stable Disease: number analyzed (Participants) | 10 | 5
  Stable Disease | 20 [2.5 to 55.6] | 25 [3.2 to 65.1]
  Progressive Disease: number analyzed (Participants) | 10 | 5
  Progressive Disease | 0 [0 to 0] | 37.5 [8.5 to 75.5]
  Not Evaluable: number analyzed (Participants) | 10 | 5
  Not Evaluable | 0 [0 to 0] | 37.5 [8.5 to 75.5]

2. Secondary Outcome: Peak Level of LMB-2 in Adult T-Cell Lymphoma
Description: The maximum analyte concentration in serum was reported using a cytotoxicity assay measuring the level of LMB-2 in the plasma and using purified LMB-2 as a standard curve.
Time Frame: First 24 hours after the dose given on Cycle 2, day 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 5
ng/mL | 602 [189 to 1072] | 484 [205 to 748]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was determined by the Kaplan Meier method beginning at the on study date and continuing until progression or last follow-up without progression. Progressive disease is assessed by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma, and is the appearance of new lesions, or an increase of 50% or greater in the sum of the product of the perpendicular diameters of the measurable lesions or persistent (at least two determinations) doubling of the peripheral blood leukemic cell count.
Time Frame: 70 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 8
Months | 11.6 [1.5 to 25.2] | 1.05 [0.23 to 1.54]
Statistical Analysis 1: Comparison: Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC vs All Other Patients; Published response duration of 15 patients with leukemic adult T cell leukemia treated with Alemtuzumab; Test type: Superiority; p < 0.0001, Kaplan Meier

4. Secondary Outcome: Overall Survival (OS)
Description: OS is the time between the first day of treatment to the day of disease progression. Progressive disease is assessed by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma, and is the appearance of new lesions, or an increase of 50% or greater in the sum of the product of the perpendicular diameters of the measurable lesions or persistent (at least two determinations) doubling of the peripheral blood leukemic cell count.
Time Frame: 70 months
Population: One participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 7
Months | 18.6 [2.3 to 53.0] | 3.75 [1.3 to 16.0]

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 7 years and 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 8
Participants | 10 | 8

6. Secondary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT is a grade II-IV LMB-2 or fludarabine and cyclophosphamide (FC)-related toxicity, except vascular leak syndrome, alopecia, grade II-III allergic reaction with asymptomatic bronchospasm or urticarial is considered DLT. Grade III aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, and fever are not considered DLT. Grade IV creatine phosphokinase associated with any other DLT or not resolving to <grade II within 2 weeks is considered DLT. Hematologic toxicity is not considered DLT unless it fails to resolve to <grade 2 or baseline by day 18 after cycle 1 or after day 25 after cycles 2-7. DLT from hepatotoxicity, creatine phosphokinase, and vascular leak syndrome is assumed from LMB-2, and hematologic toxicity from fludarabine and cyclophosphamide. Grade III proteinuria lasting <2 weeks after the last dose of LMB-2 is not considered DLT, and needs to resolve to grade 0-2 prior to retreatment.
Time Frame: 30 days after last dose of LMB2
Measure: Count of Participants; unit: Participants
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

7. Secondary Outcome: Soluble Cluster of Differentiation 25 (sCD25) Between Responders and Nonresponders
Description: Tumor tissue, including lymph node or skin biopsies was examined and analysis performed by flow cytometry to determine the amount of cancer cells in the body by measuring proteins which fall off cancer cells and go into the blood.
Time Frame: First 24 hours after the dose given on Cycle 2, day 1
Population: The number 8 represents the number of responders in the Arm/Group and the number 2 represents the number of non-responders in the Arm/Group.
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 8
pg/ml
  Soluble CD25, lowest post-treatment (nadir) value | 1094 [0 to 113000] | 34591 [5198 to 319000]
  Median sCD25 Nadir for responders: number analyzed (Participants) | 8 | 0
  Median sCD25 Nadir for responders | 1082 [0 to 5999] |
  Median sCD25 Nadir for non-responders: number analyzed (Participants) | 2 | 8
  Median sCD25 Nadir for non-responders | 70713 [28425 to 113000] | 34591 [5198 to 319000]
  Median sCD25 PRE-treatment for responders: number analyzed (Participants) | 8 | 0
  Median sCD25 PRE-treatment for responders | 31893 [3163 to 190000] |
  Median sCD25 PRE-treatment for non-responders: number analyzed (Participants) | 2 | 8
  Median sCD25 PRE-treatment for non-responders | 66419 [5838 to 127000] | 17079 [3668 to 122000]

8. Secondary Outcome: Area Under the Plasma Concentration (AUC) - LMB2
Description: AUC is a measure of the plasma concentration of drug over time. It is used to characterize drug absorption. Plasma levels were analyzed by cytotoxicity assay.
Time Frame: First 24 hours after the dose given on Cycle 2, day 1
Population: Three participants were non-evaluable. One participant withdrew due to inability to receive second cycle, which was the first cycle containing LMB-2. One participant had progressive disease before first cycle of LMB2, and one participant had progressive disease after first cycle of LMB2
Measure: Median (Full Range); unit: µg/-min/mL
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 5
µg/-min/mL | 161 [53.5 to 244] | 144 [49.8 to 205]

9. Secondary Outcome: Post Treatment Effects of LMB-2 + Fludarabine and Cyclophosphamide (FC) on Normal B and T Cell Subsets by Flow Cytometry
Description: Peripheral blood was obtained and analyzed by flow cytometry.
Time Frame: First 24 hours after the dose given on Cycle 2, day 1
Population: One patient did not have flow cytometry measuring it.
Measure: Median (Full Range); unit: Cells/µL
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 8
Cells/µL
  Normal T-cells | 28 [6 to 87] | 23.5 [1 to 156]
  Normal CD4+ cells: number analyzed (Participants) | 10 | 7
  Normal CD4+ cells | 99.5 [4 to 427] | 186 [1 to 3818]
  Normal CD8+ cells | 28 [6 to 87] | 23.5 [1 to 156]
  Normal B-cells | 8 [0 to 119] | 0.5 [0 to 11]

10. Secondary Outcome: Percentage of Patients Who Developed Neutralizing Antibodies After One or More Cycles of LMB-2
Description: Blood was drawn prior to each cycle of LMB-2 to determine if the level, >75% neutralization of 1000ng/ml of LMB-2 of neutralizing antibodies is too high to give additional LMB-2. Analysis was performed by cytotoxicity assay.
Time Frame: First 24 hours after the dose given on Cycle 2, day 1
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 4
percentage of participants | 40 [3.1 to 77] | 0 [0 to 0]

11. Secondary Outcome: Duration of Response (Complete Response + Partial Response)
Description: Duration of response is defined as a response lasting for at least 4 weeks but >8 weeks and is assessed by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma. Complete remission (CR) is complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related symptoms if present before therapy and normalization of those biochemical abnormalities definitely assignable to the lymphoma. Partial response is reduction by ≥50% of leukemia cell count or ≥50% reduction in the size of all measurable lesions, and no increase in size of any measurable or evaluable lesion or appearance of new lesion.
Time Frame: 69 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 8
Weeks | 69.6 [8 to 263] | 0 [0 to 0]

12. Secondary Outcome: Plasma Clearance (CL) of LMB-2
Description: Dilutions of patient plasma was tested by cytotoxicity assays to determine plasma clearance of LMB-2.The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: First 24 hours after the dose given on Cycle 2, day 1
Population: as for outcome 8
Measure: Median (Full Range); unit: mL/min
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 5
mL/min | 109 [10.9 to 134] | 101 [13.5 to 191]

13. Secondary Outcome: Volume of Distribution of LMB-2
Description: Dilutions of patient plasma were tested by cytotoxicity assays to determine volume of distribution of LMB-2. Volume distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. This was measured during the first 24 hours after administration of the dose on cycle 2 day 1.
Time Frame: 24 hours
Population: as for outcome 8
Measure: Median (Full Range); unit: Liters
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 5
Liters | 49.6 [3.3 to 313] | 26.6 [4.89 to 133]

14. Secondary Outcome: Half Life (t1/2) of LMB-2
Description: Dilutions of patient plasma was tested by cytotoxicity assays to determine half life. Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: First 24 hours after the dose given on Cycle 2, day 1
Population: as for outcome 8
Measure: Median (Full Range); unit: min
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
Number analyzed (Participants) | 10 | 5
min | 360 [105 to 542] | 251 [91.1 to 484]

15. Secondary Outcome: Count of Participants With Grades 3-5 Adverse Events of > 1 Adult T-Cell Leukemia (ATL) Patients Treated With 20+200, 25+250, and 30+300 mg/m^2 LMB-2/Fludarabine and Cyclophosphamide
Description: Adverse events is assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 3 (mild), Grade 4 (life threatening) and Grade 5 (death).
Time Frame: 7 years and 12 days
Population: Data for this outcome measure is reported as in the publication noted in the References module.
Measure: Count of Participants; unit: Participants
Groups:
- Fludarabine and Cyclophosphamide: 20 + 200mg/m^2: Patients CF15, CF16, and CF17. Patient CF15 did not receive LMB-2, others received 40 µg/kg.
- Fludarabine and Cyclophosphamide: 25 + 250mg/m^2: All other patients, including CF18 and CF01 who did not receive LMB2. Patients CF02 and CF03 and CF04 received LMB-2 30 µg/kg, others 40 µg/kg.
- Fludarabine and Cyclophosphamide: 30 + 300mg/m^2: Patients CF08 and CF09, both received LMB-2 40 µg/kg
Arm/Group | Fludarabine and Cyclophosphamide: 20 + 200mg/m^2 | Fludarabine and Cyclophosphamide: 25 + 250mg/m^2 | Fludarabine and Cyclophosphamide: 30 + 300mg/m^2
Number analyzed (Participants) | 3 | 12 | 2
Participants
  Neutropenia | 2 | 10 | 2
  Nausea/vomiting/anorexia | 2 | 10 | 2
  Fever/chills | 1 | 10 | 1
  Leukopenia/lymphopenia | 1 | 9 | 2
  Transaminases | 3 | 8 | 1
  Hypotension/tachycardia | 1 | 8 | 2
  Thrombocytopenia | 1 | 8 | 2
  Anemia | 0 | 9 | 1
  Myalgia/headache | 2 | 7 | 2
  Hypoalbuminemia | 2 | 6 | 1
  Hematuria | 1 | 5 | 1
  Proteinuria | 0 | 7 | 0
  Fatigue/dizziness | 1 | 4 | 2
  Edema | 0 | 6 | 0
  Abdominal pain | 0 | 5 | 0
  Diarrhea | 1 | 3 | 0
  Creatine phosphokinase (CPK) | 0 | 4 | 0
  Mucositis | 0 | 3 | 1
  Hypomagnesemia | 0 | 3 | 0
  Bilirubin | 1 | 2 | 0
  Alkaline phosphatase/gamma-glutamyl transferase | 0 | 3 | 0
  Pneumonitis | 0 | 3 | 0
  Low cluster of differentiation 4 (CD4) count | 1 | 1 | 1
  Lipase | 0 | 3 | 0
  Bladder infection | 0 | 2 | 0
  Dyspnea | 0 | 2 | 0
  Prothrombin time | 1 | 1 | 0
  Pruritis | 1 | 0 | 1

16. Secondary Outcome: Count of Participants With Adverse Events Attributed At Least Possibly to Patients Treated With Fludarabine and Cyclophosphamide Dose Levels 20+200, 25+250, and 30+300 mg/m^2
Description: Adverse events is assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 7 years and 12 days
Population: *Grade 5 (death) event. Data for this outcome measure is reported as in the publication noted in the References module.
Measure: Count of Participants; unit: Participants
Groups:
- 3Fludarabine and Cyclophosphamide: 0 + 300mg/m^2: Patients CF08 and CF09, both received LMB-2 40 µg/kg
Arm/Group | Fludarabine and Cyclophosphamide: 20 + 200mg/m^2 | Fludarabine and Cyclophosphamide: 25 + 250mg/m^2 | 3Fludarabine and Cyclophosphamide: 0 + 300mg/m^2
Number analyzed (Participants) | 3 | 12 | 2
Participants
  Neutropenia | 1 | 9 | 2
  Leukopenia/lymphopenia | 1 | 9 | 2
  Anemia | 0 | 8 | 0
  Transaminases | 1 | 4 | 0
  Thrombocytopenia | 0 | 5 | 1
  Fever/chills | 0 | 3 | 1
  Pneumonitis | 0 | 3 | 0
  Low cluster of differentiation 4 (CD4) count | 1 | 1 | 1
  Hypotension/tachycardia | 0 | 2 | 0
  Rectal hemorrhage | 0 | 1 | 0
  Bilirubin | 0 | 1 | 0
  Dysuria | 0 | 1 | 0
  Bladder infection | 0 | 1 | 0
  Hypoxia | 0 | 1 | 0
  Proteinuria | 0 | 1 | 0
  Sepsis* | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 7 years and 12 days
Arm/Group | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC | All Other Patients
All-Cause Mortality (participants affected / at risk) | 8/10 | 6/8
Serious Adverse Events (participants affected / at risk) | 7/10 | 6/8
Other Adverse Events (participants affected / at risk) | 10/10 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC (N=10) | All Other Patients (N=8)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Death
Death related to disease (General disorders) | 7 (7) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leukemic Patients Receiving LMB-2 & At Least 25+250 mg/m^2 FC (N=10) | All Other Patients (N=8)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (20) | 2 (2)
Alkaline phosphatase increased (Investigations) | 7 (9) | 3 (4)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (108) | 5 (16)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (44) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 5 (10) | 3 (3)
Blood and lymphatic system disorders - Other,Prothrombin time prolonged (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 2 (6) | 1 (2)
CPK increased (Investigations) | 5 (6) | 3 (4)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Chills (General disorders) | 5 (10) | 1 (1)
Confusion (Psychiatric disorders) | 2 (3) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (10) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 4 (8) | 0 (0)
Edema limbs (General disorders) | 7 (12) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 2 (3) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (7) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (6) | 1 (1)
Fever (General disorders) | 10 (23) | 7 (7)
Fibrinogen decreased (Investigations) | 2 (3) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0)
GGT increased (Investigations) | 4 (5) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Haptoglobin decreased (Investigations) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 7 (16) | 3 (5)
Hematuria (Renal and urinary disorders) | 5 (10) | 2 (2)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (9) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 3 (9) | 2 (2)
Hypertension (Vascular disorders) | 1 (3) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (36) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (39) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (52) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (22) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 8 (33) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (24) | 2 (2)
Hypotension (Vascular disorders) | 9 (15) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Infections and infestations - Other, CMV reaction (Infections and infestations) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Investigations - Other, Bicarbonate, low; Bicarbonate, serum-low (Investigations) | 1 (3) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 3 (3)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 9 (136) | 5 (22)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, Bicarbonate, Low (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 4 (4) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (16) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (23) | 6 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (83) | 5 (23)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (12) | 3 (4)
Papilledema (Eye disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 10 (100) | 4 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (7) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (9) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 4 (5) | 2 (2)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (6) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other,Dermatology/Skin: Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (7) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 3 (3) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (17) | 3 (6)
Weight gain (Investigations) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 8 (155) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 5 (22)
Infections and Infestations - Other, Bladder (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, tooth infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT00924170/Prot_SAP_005.pdf
  • Informed Consent Form: Eligibility Screening (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT00924170/ICF_002.pdf
  • Informed Consent Form: Standard (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT00924170/ICF_006.pdf